CLINICAL TRIAL: NCT00001096
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of HIV-1 MN rsgp120 and Bivalent AIDSVAX B/E (HIV-1 MN rgp120/A244 rgp120) in Combination With QS-21 With or Without Alum in Healthy HIV-1 Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 036; 10585 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV Antibodies; HIV Antigens; HIV-1; Adjuvants, Immunologic; AIDS Vaccines; T-Lymphocytes, Cytotoxic; HIV Seronegativity; HIV Envelope Protein gp120; Alum Compounds; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — saponin QA-21V1

INTERVENTIONS:
Biological: MN rgp120/HIV-1 and A244 rgp120/HIV-1
Biological: QS-21
Biological: rgp120/HIV-1MN

SUMMARY:
To assess the safety and immune response to two experimental vaccines when formulated with QS-21 or QS-21 plus alum. To determine whether the new preparation of QS-21 in polysorbate 80 is less reactogenic than the QS-21 formulation used in AVEG Protocols 016, 016A, and 016B. To examine whether QS-21 is immunologically equivalent to that used in 16B. To determine if QS-21, when given with low doses of antigen, induces measurable HIV-1-specific CTL activity. To evaluate if the QS-21 dose-sparing effect extends to an antigen dose of 0.5 micrograms. To determine if the bivalent vaccine gives responses equivalent to the monovalent product or if a broadening of the HIV-1-specific binding and neutralizing antibody responses occurs.

An effective vaccine to prevent HIV-1 infection may need to generate diverse and multifaceted immunologic responses. Required parts of the immune response may include: humoral antibodies, which broadly neutralize non-syncytium-inducing strains of HIV-1; T cell help provided by both CD4 and CD8 positive subsets; and a class I-restricted cytotoxic lymphocyte response. Other effector responses, such as the generation of antibody-dependent cellular cytotoxicity, cytokines, chemokines, or other antiviral factors may also be critical in mounting protective immunity. Given the lack of a surrogate immunologic marker, the most practical approach for possible efficacy trials would be to evaluate a candidate vaccine that elicits as many of these responses as possible.

DETAILED DESCRIPTION:
An effective vaccine to prevent HIV-1 infection may need to generate diverse and multifaceted immunologic responses. Required parts of the immune response may include: humoral antibodies, which broadly neutralize non-syncytium-inducing strains of HIV-1; T cell help provided by both CD4 and CD8 positive subsets; and a class I-restricted cytotoxic lymphocyte response. Other effector responses, such as the generation of antibody-dependent cellular cytotoxicity, cytokines, chemokines, or other antiviral factors may also be critical in mounting protective immunity. Given the lack of a surrogate immunologic marker, the most practical approach for possible efficacy trials would be to evaluate a candidate vaccine that elicits as many of these responses as possible.

Volunteers in each of 5 groups receive vaccine or placebo by intramuscular injection at Months 0, 1, and 6. All patients receive one of two doses of QS-21 along with vaccine or placebo and some groups receive alum as follows:

Group 1: low-dose MN rsgp120/HIV-1 plus QS-21 (13 volunteers). Group 2: high-dose MN rsgp120/HIV-1 plus QS-21 (13 volunteers). Group 3: AIDSVAX B/E (injection contains each of the two vaccine components, HIV-1 MN rgp120 and A244 rgp120/HIV-1) plus QS-21 plus alum (13 volunteers).

Group 4: high-dose MN rgp120/HIV-1 plus QS-21 plus alum (13 volunteers). Group 5: placebo plus QS-21 (8 volunteers). Volunteers will be closely monitored after each immunization and followed for a minimum of 12 months after the initial immunization.

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Negative ELISA for HIV within 8 weeks prior to immunization.
* CD4 count greater than or equal to 400 cells/mm3.
* Normal history and physical examination. [Refer to Laboratory values for additional requirements.]

Exclusion Criteria

Co-existing Condition:

Volunteers with the following conditions or symptoms are excluded:

* Medical or psychiatric conditions or occupational responsibilities which preclude subject compliance with the protocol.
* Recent suicidal ideation or psychosis.
* Active syphilis. NOTE: If the serology is documented to be a false positive or due to a remote (greater than 6 months) treated infection, the volunteer is eligible.
* Active tuberculosis. NOTE: Volunteers with a positive PPD and a normal chest x-ray showing no evidence of TB and not requiring INH therapy are eligible.
* Positive for hepatitis B surface antigen.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* History of cancer unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure.
* History of suicide attempts, recent suicidal ideation, or past or present psychosis.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance requiring hospitalization or emergency medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* History of reaction to thimerosal.

Prior Medication:

Excluded:

* Live attenuated vaccine within 60 days of study. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 2 weeks away from HIV immunizations.
* Experimental agents within 30 days prior to study.
* HIV-1 vaccines or placebo as part of a previous HIV vaccine trial.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin in the past 6 months.
* Experimental agents within 30 days prior to study.

Risk Behavior:

Excluded:

* Volunteers with an identifiable higher- or intermediate-risk sexual behavior for HIV infection (i.e., AVEG Risk Groups C or D ).
* History of intravenous drug use within 12 months prior to enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Evans, Study Chair
Locations (4):
- United States (4):
  - JHU AVEG, Baltimore, Maryland
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Evans TG, McElrath MJ, Matthews T, Montefiori D, Weinhold K, Wolff M, Keefer MC, Kallas EG, Corey L, Gorse GJ, Belshe R, Graham BS, Spearman PW, Schwartz D, Mulligan MJ, Goepfert P, Fast P, Berman P, Powell M, Francis D; NIAID AIDS Vaccine Evaluation Group. QS-21 promotes an adjuvant effect allowing for reduced antigen dose during HIV-1 envelope subunit immunization in humans. Vaccine. 2001 Feb 28;19(15-16):2080-91. doi: 10.1016/s0264-410x(00)00415-1. PMID 11228380